CLINICAL TRIAL: NCT03650699
Title: Rehabilitation of Head and Neck Cancer Patients With Biofeedback Training to Improve Speaking and Eating in Public
Brief Title: Biofeedback Rehabilitation to Improve Speaking and Eating in Public
Acronym: Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-5105
Record Dates: First submitted 2018-05-29; First posted 2018-08-29 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
Keywords: Oral Cavity Squamous Cell Carcinoma; Biofeedback; Rehabilitation; Head and Neck Cancer; electropalatography; EPG
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Directed Tongue Strengthening Rehab (Experimental): 8 sessions of self-directed tongue strengthening exercises followed by 8 sessions of electropalatography biofeedback training.
  Assessments will be taken during the beginning, middle, and end of each study arm.
  Interventions: Device: Electropalatography Biofeedback Training
- SLP Directed Face-to-Face Rehab (Experimental): 8 sessions of SLP-directed face-to-face rehabilitation program followed by 8 sessions of electropalatography biofeedback training.
  Assessments will be taken during the beginning, middle, and end of each study arm.
  Interventions: Device: Electropalatography Biofeedback Training

INTERVENTIONS:
Device: Electropalatography Biofeedback Training — The study agent is electropalatography (EPG). The LinguaGraph EPG device is a biofeedback technology that creates a digital visualization of tongue function during speech. The visualization is accomplished by a custom made mouthpiece that fits over the hard palate with 62 sensors that capture tongue position. The information from the sensors in the mouthpiece, as well as the audio output, is processed in an EPG Unit that converts the information from mouthpiece to a visual representation on a computer screen. The visual information with respect to tongue position can be used to provide biofeedback training.The computer can be used in the clinic during a patient visit or it can be seen over the internet with the patient at home and the speech and language pathologist at the clinic.

SUMMARY:
Tongue cancer requires resection and reconstruction that can leave patients disabled with respect to speaking and eating. Impairment of tongue function can have significant impact on social interaction and employment. To try and improve speaking and eating in public, the team at the University Health Network is going to use a special device that is designed to help the patient rehabilitate after tongue cancer treatment.

The research part of this study is to use a special mouthpiece or mold that is like a partial plate for upper dentures that will fit on the roof of the mouth. This mold is embedded with 62 sensors that will allow patients to visualize their tongue position during speech. With the help of a speech therapist, patients can learn different tongue positions important speaking and eating. This whole process is called biofeedback. The visualization of the tongue gives the patient the flexibility to practice at home to and learn different tongue positions important to eating and speaking. In addition, the device will provide the speech pathologist with an opportunity for easier and more precise assessment of the patient's progress which can reduce the need for visits to the hospital. The investigators expect the biofeedback training to improve the patient's speaking and eating.

The study hypothesis is that the biofeedback device will improve speech intelligibility, eating in public, speaking in public, and oral intake scores.

DETAILED DESCRIPTION:
Subjects will be enrolled in either arm of the study for duration of 4 months. Patients that are randomized into study arm 1 will come to the clinic for Speech Language Pathologist (SLP) directed face-to-face rehabilitation for a period of 2 months. The patients will then transition to participate in weekly face-to-face Electropalatography (EPG) biofeedback training. The EPG biofeedback will be used for 2 months. Patients that are randomized into study arm 2 will first undergo a self-directed tongue strengthening program (oral exercises) for a period of 2 months and then transition into EPG biofeedback training.

Although randomization will be used, this is a nonstandard trial because all patients will receive biofeedback EPG. Patients from both study arms will receive biofeedback training after undergoing an SLP directed face-to-face rehabilitation program versus a self-directed tongue strengthening program (oral exercises). The SLP directed face-to-face rehabilitation program or self-directed tongue strengthening program will be initiated at least 2 weeks post-surgery. If the patient is treated with adjuvant radiation, the patient will take a self-directed biofeedback holiday with a target of restarting at least 2 after the completion of adjuvant treatment.

This design was chosen because there is equipoise with respect to the efficacy of the intervention and uncertainty with respect to whether the intervention is most valuable following an SLP directed face-to-face rehabilitation program versus a self-directed tongue strengthening program. The design offers all patients the opportunity to participate in the intervention. This approach will also allow us to analyze between subject change and within subject change.

The A.I.D.S assessment has been in place for approximately 50 years. The mean A.I.D.S. efficiency score (95%CI) in the current pilot study (n=16) is 0.54 (46.0, 62.3). With 33 patients in each group, there will be over 80% power to detect a 10% difference in the speech efficiency score even under the condition that there may be low (rho<0.1) correlation within subject. Higher correlation within subject on the various scores would serve to increase the efficiency of the analysis.

Bivariate comparison will be made between the arms with respect to the primary and secondary outcome variables at each time point.

Linear mixed model will be used to account for multiple measures at multiple time points. The first step will be to compare arms with respect to the primary and secondary outcome variables. For those tests that are significant a backward selected regression will be performed to control for confounders and to look for important effect modifier variables. Variables related to rehabilitation participation will be modeled in the backward selected regression.

ELIGIBILITY:
Inclusion Criteria:

* Oral cavity carcinoma involving the tongue or floor of the mouth
* Primary surgical treatment or/
* Primary surgical treatment with adjuvant radiation therapy or/
* Salvage surgical treatment
* At least 2 weeks post treatment

Exclusion Criteria:

* Anatomic palate abnormality that precludes fitting a mouthpiece
* Cognitively unable to participate in biofeedback
* Persistent Cancer
* Does not speak English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Percent Intelligibility of Speech Over 4 Months | Administered at 0, 2, and 4 months
  Change in percent intelligibility is measured using Assessment of Intelligibility of Dysarthric Speech (AIDS). Assessment of Intelligibility of Dysarthric Speech (AIDS) is a validated tool that is used in this outcome to measure intelligibility as compared with normal subjects for quantifying single-word intelligibility and sentence intelligibility.
Change in Rate of Intelligible Speech Over 4 Months | Administered at 0, 2, and 4 months
  Change in intelligibility rate is also measured using Assessment of Intelligibility of Dysarthric Speech (AIDS). Assessment of Intelligibility of Dysarthric Speech (AIDS) is a validated tool that is used in this outcome to measure speed of language as compared with normal subjects for quantifying speaking rate.
Change in Speech Acceptability Over 4 Months | Administered at 0, 2, and 4 months
  Assessment of Speech Acceptability is a qualitative measure of "conversational understandability" of language as compared with normal subjects. Subjects will be given 6-word sentences to read where five naïve listeners will evaluate the speakers' speech acceptability on a scale of 4. This is a subsection of the AIDS test.
Change in Speech and Swallowing Over 4 Months | Administered at 0, 2, and 4 months
  This is a disease specific, 6-item, administered questionnaire to evaluate post-treatment speech and swallowing ability measure will provide critical data on the socialization of the patient as it relates to speaking and eating.

SECONDARY OUTCOMES:
Change in Patient Satisfaction of EPG Biofeedback Over 4 Months | Administered time 0, 2, and 4 months
  The patient will be given a self-administered questionnaire to assess satisfaction and adoption of biofeedback.
Difference in Cost for Intervention versus Standard of Care Over Time | Weekly, Up to 16 Weeks
  Hospital, personnel and patient cost will be collected. SLP time will be recorded on time sheets. The fuel and parking cost will be imputed based on the first 3 numbers of the postal code.

OTHER OUTCOMES:
Measure of Obliteration using Oral Volume Assessment Tool (OVAT) | Administered at 0, 2, and 4 months
  Obliteration of the oral cavity is defined as the ability of the tongue volume to obliterate the oral cavity so that there is space between the tongue and the hard and soft palate. Obliteration is measured using the Oral Volume Assessment Tool (OVAT) which is a measure of displacement. This is an important mechanism of bolus propulsion during the oral phase of swallowing.
Measure of Tongue Protrusion | Administered at 0, 2, and 4 months
  Protrusion of the tongue is defined as the distance the tongue can be extended beyond the central mandibular incisors measured in millimeters. This is important for the finger function of the tongue.
Measure of Tongue Elevation | Administered at 0, 2, and 4 months
  Elevation of the tongue is defined as distance the tongue can be moved superiorly above the central mandibular incisors measured in millimeters. The goal is to obtain premaxillary contact.
Fiberoptic Endoscopic Evaluation of Swallow (FEES) | Administered time 0, 2, and 4 months
  FEES is an assessment that involves placing a flexible endoscope transnasally to obtain a superior view of the pharynx and larynx. The purpose is to evaluate structure & function of the upper aerodigestive tract. This assessment enables visualization nasopharynx, base of the tongue, oropharynx, hypopharynx, and larynx. FEES is used for assessment of retained secretions and retained food consistencies. It is useful for assessing airway protection as it relates to swallowing function. After assessment, FEES is useful for evaluation of the effectiveness of compensatory techniques (postures, maneuvers, bolus modifications) for improving swallowing safety and efficiency. This is a standard of care assessment but is not routinely performed on all OCSCC patients. The surgeon/SLP will use FEES to look at swallowing function and the effectiveness of rehabilitation.
Clinical Speech and Language Assessment | Weekly, Up to 16 weeks
  This is documentation of data that would appear in a clinical speech and language consultation. There are parts of the assessment that cannot be performed if the patient does not return to the hospital and the consultation is performed with a video link. These sections of the assessment will be marked "missing data" on the data sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Chepeha, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada